CLINICAL TRIAL: NCT02468882
Title: Does Watercress Intake Have an Impact on Cancer Patients Outcomes: a Randomized Longitudinal Trial
Brief Title: Does Watercress Intake Have an Impact on Cancer Patients Outcomes: a Longitudinal Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Paula Ravasco, Principal Investigator, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ULisbon
Record Dates: First submitted 2015-05-21; First posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Long-term Effects Secondary to Cancer Therapy in Adults
Keywords: Breast cancer; Radiotherapy; Toxicity; Outcomes; Watercress
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Watercress will be tested in its natural form as a food item that will supplement the usual diet, via the prescription of watercress as whole food added daily to the usual diet. The intervention group will be asked to consume 100 grams of watercress per day, in addition to their usual diet for the total time of RT treatment. These 100 grams of watercress per day will allow the achievement of the daily "therapeutic" dose.
  Interventions: Dietary Supplement: Watercress
- Control group (No Intervention): The control group will receive the standard of care, thus will maintain their ad libitum diet.

INTERVENTIONS:
Dietary Supplement: Watercress — 100g of watercress daily during radiation therapy
  Arms: Intervention group

SUMMARY:
Population studies associate a higher intake of cruciferous vegetables with a reduced risk of cancer. Studies identified PEITC and several active isothiocyanates in watercress extract that may have significant anticarcinogenic activity. Potential anticarcinogenic mechanisms include: preventing carcinogen activation by inhibiting phase I enzymes such as cytochrome P450s, by increasing cells' resistance through detoxification/antioxidant enzymes, by inhibiting cell cycle progression and/or by inducing apoptosis.

These findings are justifiably interesting for the primary care setting and cancer primary prevention. Yet, these cellular effects of watercress supplementation may further prove useful in the modulation of cancer progression and disease recurrence. The present clinical trial of nutritional supplementation in cancer, intends to further explore the effects of therapeutic diets supplemented with nutraceuticals via watercress that may prove useful in DNA damage modulation, as well as in the global disease prognosis.

DETAILED DESCRIPTION:
The relation between cancer and nutrition has been well established; cancer builds upon damage to cellular DNA resulting from carcinogenic environmental factors, in which nutrition plays a major role. Many diet and lifestyle factors can influence the development of cancer, a disease expected to affect worldwide more than 1 in 3 people. Population studies associate a higher intake of cruciferous vegetables with a reduced risk of cancers at several locations. In 1977, a study in laboratory animals showed the potential effect of phenylethyl isothiocyanate (PEITC) to inhibit carcinogenesis. Recent studies identified several active isothiocyanates in watercress extract that may have more significant anticarcinogenic activity than PEITC alone. Potential anticarcinogenic mechanisms include: preventing carcinogen activation by inhibiting phase I enzymes such as cytochrome P450s, by increasing cells' resistance through detoxification/antioxidant enzymes; e.g. phase II enzymes (quinone reductase, glutathione S-transferases, UDP glucuronosyltransferases);, by inhibiting cell cycle progression and/or by inducing apoptosis.

Several watercress components have antigenotoxic effects in vitro resulting in reduced DNA damage and have anti-proliferative effects. These components include flavonols such as quercetin, hydroxycinnamic acids such as ferulic acid and p-coumaric acid. In HT29 colon cancer cells, an extract of watercress juice was associated with inhibition of the three stages of carcinogenesis: initiation, proliferation and metastasis. In MDA-MB-23 human breast cancer cells, watercress extract inhibited metalloproteinase-9 activity, thus suppressing the invasive potential of cancer cells. In breast cancer, epidemiological studies suggest that cruciferous vegetables may reduce cancer incidence. In animal studies, a 9-week PEITC-NAC supplemented diet vs a non-supplemented diet was significantly associated with reduction in tumour size and weight.

A recognised mechanism by which PEITC inhibits the growth and survival of established cancer cells is through the inhibition of angiogenesis. A study explored the impact of PEITC on a specific pathway central to angiogenesis by exposing human MCF7 breast cancer cells to PEITC and measuring hypoxia inducible factor (HIF) signaling activity. PEITC was shown as an effective inhibitor of HIF activity which may contribute to its anti-angiogenic and anti-cancer properties. A follow up to this experiment demonstrated that, similar to PEITC, crude watercress extracts inhibited cancer cell growth and HIF activity in vitro. Furthermore 6 to 8 hours after a significant amount dietary intake of watercress by four healthy participants, peripheral blood cells demonstrated significantly reduced HIF signalling activity, suggesting that dietary intake of watercress may be sufficient to modulate this potential anti-cancer pathway.

Of further relevance, a blind, randomized crossover study was carried out in 60 healthy volunteers instructed to consume one pack (85g) of raw watercress daily for 8 weeks. Compared to the control phase, watercress supplementation increased lymphocytes' DNA resistance to free radicals, thus reducing DNA damage. The hypothesis set out was that watercress may reduce cancer risk via decreased damage to DNA and possible effects on antioxidant status by increasing levels of plasma carotenoids.

These findings are justifiably interesting for the primary care setting and cancer primary prevention. Yet, these cellular effects of watercress supplementation may further prove useful in the modulation of cancer progression and disease recurrence, a not yet explored area. Of note, that the role of nutrition intervention in medium and long term outcomes in cancer has been demonstrated. It is today acknowledged as grade A evidence that individualized nutritional counseling and education plays a central role in improving long-term outcomes in cancer, by prolonging survival, reducing late RT toxicity and improving QoL. The present clinical trial of nutritional supplementation in cancer, intends to further explore the effects of therapeutic diets supplemented with nutraceuticals via watercress that may prove useful in DNA damage modulation, as well as in the global disease prognosis.

ELIGIBILITY:
Inclusion Criteria:

* adult breast cancer female patients consecutively referred for primary radiotherapy with curative intent

Exclusion Criteria:

* pregnancy
* cognitive impairment
* uncooperative or
* patients with any implantable electronic device (e.g. pacemaker) or internal metal material preventing BIA phase angle assessment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Cell phase angle | Change from baseline at up to 6 weeks
  as an indirect measure of cell membrane integrity, function and metabolism
body composition | Change from baseline at up to 6 weeks
  assessed by tetrapolar multifrequency Bioimpedance Analysis (BIA) and CT scan images; CT scans analysis will be performed in collaboration with expert groups
treatments' toxicity and symptoms | up to 6 weeks
  Assessed by the RTOG Common Toxicity Criteria, developed by the Eastern Cooperative Oncology Group (RTOG)
RT induced skin dermitis | up to 6weeks
  Evaluated by a radiation oncologist, using a validated toxicity scale
Quality of Life (QoL) | Change from baseline at up to 6 weeks
  will be assessed by the European Organisation for Research and Treatment of Cancer (EORTC-QLQ C30), validated for Oncology
DNA damage | Change from baseline at up to 6 weeks
  DNA damage assessment by Comet assay in lymphocytes has been used extensively as a surrogate biomarker to measure exposure to genotoxic agents and assess cancer risk in human studies by us and others. biological samples will comprise serum or plasma (1 mL) prepared from blood samples collected in Heparin tubes and urine (1 mL). Metabolomic profiles will be measured on a 700 MHz 1H NMR spectrometer equipped with a cryo-probe for enhanced sensitivity. 1H NMR spectroscopy: high throughput metabolic phenotyping is a powerful approach for characterising biochemical signatures of biological samples. We will couple high-resolution 1H NMR spectroscopy and mathematical modelling approaches to determine the metabolic profile in biological samples from patients.
Metabolomic profile | Change from baseline at up to 6 weeks
  Metabolomics simultaneously measures thousands of low molecular weight metabolites providing holistic information on the biochemical status of the body. Previous metabolomic studies have identified cancer-associated perturbations in the metabolic phenotypes of patients. This study will explore the ability of watercress to improve the restorative effects of radiotherapy in breast cancer patients on the metabolic status towards a healthy phenotype
Nutritional status | Change from baseline at up to 6 weeks
  assessed by the method Patient-Generated Subjective Global Assessment, specific and validated for Oncology
Dietary intake | Change from baseline at up to 6 weeks
  Will derive from a diet history and a 24-hour-recall food questionnaire. The software Dietplan6 (Forestfield Software Ltd 2013®, Horsham, UK) will analyze the nutrient content of foods consumed
Carotenoids and flavonoids | Change from baseline at up to 6 weeks
  The plasma samples analysis will also include the measurement of carotenoids and flavonoids, which are present in watercress, and are related with antigenotoxic effects in vitro and have anti-proliferative effects, as demonstrated in several studies. Urine samples analysis will allow the measurement of flavonoids.

SECONDARY OUTCOMES:
Cell phase angle 2 | change from 3 months at 3 years
  as an indirect measure of cell membrane integrity, function and metabolism
body composition 2 | change from 3 months at 3 years
  assessed by tetrapolar multifrequency Bioimpedance Analysis (BIA)
Quality of Life 2 (QoL2) | change from 3 months at 3 years
  will be assessed by the European Organisation for Research and Treatment of Cancer (EORTC-QLQ C30), validated for Oncology
Metabolomic profile 2 | change from 3 months at 3 years
  Metabolomics simultaneously measures thousands of low molecular weight metabolites providing holistic information on the biochemical status of the body. Previous metabolomic studies have identified cancer-associated perturbations in the metabolic phenotypes of patients. This study will explore the ability of watercress to improve the restorative effects of radiotherapy in breast cancer patients on the metabolic status towards a healthy phenotype
Nutritional status 2 | change from 3 months at 3 years
  assessed by the method Patient-Generated Subjective Global Assessment, specific and validated for Oncology
Dietary intake 2 | change from 3 months at 3 years
  Will derive from a diet history and a 24-hour-recall food questionnaire. The software Dietplan6 (Forestfield Software Ltd 2013®, Horsham, UK) will analyze the nutrient content of foods consumed

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Santa Maria, Lisbon, Portugal